CLINICAL TRIAL: NCT05336747
Title: Here, My Voice 2 - Voice Lessons Pilot
Brief Title: Here, My Voice 2 Voice Lessons Pilot
Acronym: HMV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Marientina Gotsis, Professor of Practice, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UP-22-00164
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hearing Loss
Keywords: cochlear implants; voice lessons
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice Lessons "Here, My Voice 2" Program (Experimental): Voice Lessons "Here, My Voice 2" Program
  Interventions: Behavioral: Voice lessons
- Voice Lessons "Here, My Voice 3" Program (Experimental): Voice Lessons "Here, My Voice 3" Program
  Interventions: Behavioral: Voice lessons

INTERVENTIONS:
Behavioral: Voice lessons — 12 x 60 minute one-on-one vocal training lessons, once weekly in person or over videoconferencing, and additional 60 min per week home training of vocal pitch control using an internet based vocal pitch app.

SUMMARY:
Active music engagement has been shown to provide unique benefits for both pediatric and adult cochlear implant (CI) users. Here, My Voice 2 (HMV 2) project will build upon the 2021 pilot program and provide personalized voice lessons to members of the hard-of-hearing (HOH) community in order to support the (re)discovery of their voice as a tool of self-expression. Over the course of 12 weeks, participants from the HOH community will partner with students from USC's Thornton School of Music to practice expressive vocal techniques in one-on-one individual lessons. At the conclusion of the lessons, HLAA will host a communal session with a recital in which each team will present what they have worked on. Data will be collected via self-assessment surveys, vocal assessment measures, and interviews at the beginning, middle, and end of the program, as well as a 3 month follow-up. This data will be quantified/coded using qualitative coding, as appropriate, and the findings will be published in relevant conferences and journals. The data will also be used to evaluate the merits of this program to improve the format in future iterations.

ELIGIBILITY:
Inclusion Criteria:

* Adults, English speaking, who experience profound hearing loss and use cochlear implants or/and hearing aids.
* Ability to use voice without discomfort and without causing any health issues.
* Ability to commit one hour a week over a 12-week period and an additional 10 min period of daily training.

Exclusion Criteria:

* People with medical conditions such as tracheostomy, which makes using voice difficult and potentially threatens their health
* People taking part in other training programs for vocal, musical or auditory skills in the same time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Change in Vocal Confidence | Change between baseline and 1 week post voice lessons
  Vocal confidence will be measured using a questionnaire developed by USC's Bionic Ear Lab researchers combined with Singing Voice Handicap Index (SVHI) to measure levels of self-esteem as well as physical and emotional experiences related to singing.
Change in Goldsmiths Musical Sophistication Index (Gold MSI) | Change between baseline and 1 week post voice lessons
  The Goldsmiths Musical Sophistication Index measures musical attitudes, behaviours, and skills
Change in Quality of Life in Neurological Disorders (Neuro-QoL) Questionnaire | Change between baseline and 1 week post voice lessons
  The specific domains assessed in Neurological Disorders (Neuro-QoL) Questionnaire will include: ability to participate in social roles and activities, positive affect and well-being, and satisfaction with social roles and activities.
Change in Auditory Skills | Change between baseline and 1 week post voice lessons
  Speech and music perceptual abilities via TeamHearing software.
Change in Vocal Skills of Audio Recordings of Participants | Change between baseline and 1 week post voice lessons
  Pitch matching, interval matching, and rhythm matching abilities will be rated automatically for accuracy by Praat speech analysis software and additional characteristics of vocal quality and singing accuracy (melodic contour, diction, tempo, tone, phrasing, and breath) will be rated by voice teachers on a Likert-type scale (0-5 with higher being more accurate).
Change in Self Esteem | Change between baseline and 1 week post voice lessons
  The Rosenberg Self Esteem Scale is a10-item self-reported questionnaire designed to measure self-esteem. It includes 10 statements related to a person's feelings of self-worth or self-acceptance. A four-point scale ranging from "strongly agree" to "strongly disagree" is used to answer the questions (Rosenberg Self-Esteem Scale, n.d). The RSES is a reliable instrument as indicated by its Guttman scale coefficient of reproducibility of 0.92, which indicates excellent internal consistency. Test-retest reliability has correlations of 0.85 and 0.88 over a 2-week period, which indicates appropriate stability. The validity of the RSES is demonstrated by its concurrent, predictive, and constructive validity using known groups. The RSES correlates significantly with other measures of self-esteem such as the Coopersmith Self-Esteem Inventory as well as with the predicted direction of measures of depression and anxiety (Rosenberg, 2006).

SECONDARY OUTCOMES:
Participation motivation, experience, and goals | Up to 14 weeks
  Semi-structured interviews will be used to assess participant motivation and quality of experience within the program. Responses will be qualitatively coded and compared from baseline to the end of the program.
Engagement of the participants | Up to 12 weeks
  Voice teachers will keep a teaching log reflecting upon participants' attendance, motivation, and engagement.These notes will be compiled and coded following the program to qualitatively track vocal progress of participants throughout the study.
Changes in Vocal Skills of Participants | Up to 12 weeks
  Voice teachers will keep a teaching log reflecting upon student progress and which techniques, vocal warm-ups, or other learning methods proved most effective during lessons. These notes will be compiled and coded following the program to qualitatively track vocal progress of participants throughout the study.
Changes in Vocal Confidence | Change between 1 week post voice lessons and 3 months post voice lessons
  Vocal confidence will be measured using a questionnaire developed by USC's Bionic Ear Lab researchers combined with Singing Voice Handicap Index (SVHI) to measure levels of self-esteem as well as physical and emotional experiences related to singing.
Change in Goldsmiths Musical Sophistication Index (Gold MSI) | Change between 1 week post voice lessons and 3 months post voice lessons
  The Goldsmiths Musical Sophistication Index measures musical attitudes, behaviours, and skills
Change in Quality of Life in Neurological Disorders (Neuro-QoL) Questionnaire | Change between 1 week post voice lessons and 3 months post voice lessons
  The specific domains assessed in Neurological Disorders (Neuro-QoL) Questionnaire will include: ability to participate in social roles and activities, positive affect and well-being, and satisfaction with social roles and activities.
Change in Auditory Skills | Change between 1 week post voice lessons and 3 months post voice lessons
  Speech and music perceptual abilities via TeamHearing software
Change in Vocal Skills of Audio Recordings of Participants | Change between 1 week post voice lessons and 3 months post voice lessons
  Pitch matching, interval matching, and rhythm matching abilities will be rated automatically for accuracy by Praat speech analysis software and additional characteristics of vocal quality and singing accuracy (melodic contour, diction, tempo, tone, phrasing, and breath) will be rated by voice teachers on a Likert-type scale (0-5 with higher being more accurate)
Change in Self Esteem | Change between 1 week post voice lessons and 3 months post voice lessons
  The Rosenberg Self Esteem Scale is a10-item self-reported questionnaire designed to measure self-esteem. It includes 10 statements related to a person's feelings of self-worth or self-acceptance. A four-point scale ranging from "strongly agree" to "strongly disagree" is used to answer the questions (Rosenberg Self-Esteem Scale, n.d). The RSES is a reliable instrument as indicated by its Guttman scale coefficient of reproducibility of 0.92, which indicates excellent internal consistency. Test-retest reliability has correlations of 0.85 and 0.88 over a 2-week period, which indicates appropriate stability. The validity of the RSES is demonstrated by its concurrent, predictive, and constructive validity using known groups. The RSES correlates significantly with other measures of self-esteem such as the Coopersmith Self-Esteem Inventory as well as with the predicted direction of measures of depression and anxiety (Rosenberg, 2006).
Changes in Music Experience UCMLQ Questionnaire | Change between baseline and 1 week post voice lessons
  University of Canterbury Music Listening Questionnaire (UCMLQ) questionnaire will measure participants music experience with Hearing Aids or/and Cochlear Implants

CONTACTS AND LOCATIONS:
Overall Officials: Juri Hwang, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No